CLINICAL TRIAL: NCT03852030
Title: Mind-Body Health in Uro-Oncology: A Randomized Controlled Trial
Brief Title: Mind-Body Health in Uro-Oncology: Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Endeavor Health (Other)
Responsible Party: Principal Investigator, David Victorson, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EH09-202
Record Dates: First submitted 2018-12-12; First posted 2019-02-22 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer; Kidney Cancer; Bladder Cancer
Keywords: prostate cancer; mindfulness; eHealth; kidney cancer; bladder cancer; caregiver
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Following participation in the 8-week course, participants will be randomized to either 4 months of: 1) weekly MBSR specific text or email messages related to course teachings, 2) weekly general/informational texts or emails about healthy living and lifestyle, or 3) no texts or emails.
Who Masked: Participant
Masking Description: Participants were not told to which weekly text messaging group they were being assigned, or about the other groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness text/email message (Experimental): Weekly MBSR specific text or email messages related to course teachings were sent.
  TYPES OF MESSAGES INCLUDED: Non-reaction; Non-Judgment; Awareness; Loving Kindness; Acceptance.
  Interventions: Behavioral: Text or email message
- Health promotion text/email message (Placebo Comparator): Weekly general/informational texts or emails about healthy living and lifestyle were sent. TYPES OF MESSAGES INCLUDED: Diet; Exercise; Sleep; Illness; Stress.
  Interventions: Behavioral: Text or email message
- No text/email message (No Intervention): No texts or emails were sent. There are no examples or descriptions for these messages, because no messages were sent to this group.

INTERVENTIONS:
Behavioral: Text or email message — Text or email messages sent to research participants
  Arms: Health promotion text/email message; Mindfulness text/email message

SUMMARY:
In this study, the researchers will examine the effects of post-mindfulness intervention email and text messages to promote maintenance of intervention effects over time in a uro-oncology sample (clinically localized prostate, kidney, and bladder cancer) of patients and spouses.

DETAILED DESCRIPTION:
Participant accrual will occur at NorthShore University HealthSystem's John and Carol Walter Center for Urological Health. During or prior to an office visit, a potential subject and possibly his/her spouse will speak with the physician or research staff to assess interest in discussing the study. All eligible participants will be enrolled into an 8-week mindfulness-based stress reduction (MBSR) course. Because the course content focuses on training in mindfulness meditation (and not cancer-specific issues), the researchers will allow for mixed cancer classes. Prior to the first class, all participants will complete baseline standardized patient reported outcomes (PROs) of health related quality of life, and undergo blood collection via finger prick. Following participation in the 8-week course, participants will complete their 8-week PRO and bio-marker assessments in a similar manner, and will be randomized to either 4 months of: 1) weekly mindfulness-specific text or email messages related to course teachings, 2) weekly general/informational texts or emails about healthy living and lifestyle, or 3) no texts or emails. PRO and bio-marker assessments will also be administered at 6 months, and PRO measures will be collected at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with clinically localized or locally advanced prostate, kidney or bladder cancer OR the spouse/significant other (married or living together ≥ 1 year) of a person with prostate, kidney or bladder cancer
* Spouses/significant others will only be included if their partners with cancer diagnoses will be participating
* 18 years old or older
* Proficient in comprehending spoken English. Proficient in reading and writing English.

Exclusion Criteria:

* Is not able to receive email or text messages
* History of diagnosed severe mental illness or hospitalization for chronic psychiatric reasons, as identified by referring physicians, such that participation in MBSR group activities would be contraindicated.
* Vision- or hearing-impaired such that ability to listen to or observe MBSR course instructions is compromised.
* Diminished cognitive skills as to render consent meaningless
* Physical debilitation such that study participation would not be feasible or would create undue hardship.
* Participation in the intervention arm of the preceding study, "Reducing Stress During Active Surveillance" EH09-202.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
change in fatigue using the PROMIS Fatigue questionnaire | baseline, 8 weeks, 6 months, 12 months
  Examine change in fatigue between the intervention arms by comparing the responses on the PROMIS Fatigue questionnaire
change in depression using the PROMIS Depression questionnaire | baseline, 8 weeks, 6 months, 12 months
  Examine change in depression between the intervention arms by comparing the responses on the PROMIS Depression questionnaire
change in anxiety using the PROMIS Anxiety questionnaire | baseline, 8 weeks, 6 months, 12 months
  Examine change in anxiety between the intervention arms by comparing the responses on the PROMIS Anxiety questionnaire
change in sleep using the PROMIS Sleep Disturbance questionnaire | baseline, 8 weeks, 6 months, 12 months
  Examine change in sleep between the intervention arms by comparing the responses on the PROMIS Sleep Disturbance questionnaire
change in physical function using the PROMIS Physical Function questionnaire | baseline, 8 weeks, 6 months, 12 months
  Examine change in physical function between the intervention arms by comparing the responses on the PROMIS Physical Function questionnaire
change in stress using the State-Based Stress Visual Analogue Scale | baseline, 8 weeks, 6 months, 12 months
  Examine change in stress between the intervention arms by comparing the responses on the State-Based Stress Visual Analogue Scale
change in mindfulness using the 5-Facet Mindfulness Sub-scales | baseline, 8 weeks, 6 months, 12 months
  Examine change in mindfulness between the intervention arms by comparing the responses on the 5-Facet Mindfulness Subscales

CONTACTS AND LOCATIONS:
Overall Officials: David E Victorson, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latini DM, Hart SL, Knight SJ, Cowan JE, Ross PL, Duchane J, Carroll PR; CaPSURE Investigators. The relationship between anxiety and time to treatment for patients with prostate cancer on surveillance. J Urol. 2007 Sep;178(3 Pt 1):826-31; discussion 831-2. doi: 10.1016/j.juro.2007.05.039. Epub 2007 Jul 16. PMID 17632144
- [Background] Mehnert A, Lehmann C, Schulte T, Koch U. Presence of symptom distress and prostate cancer-related anxiety in patients at the beginning of cancer rehabilitation. Onkologie. 2007 Nov;30(11):551-6. doi: 10.1159/000108578. Epub 2007 Oct 16. PMID 17992025
- [Background] Miller DC, Sanda MG, Dunn RL, Montie JE, Pimentel H, Sandler HM, McLaughlin WP, Wei JT. Long-term outcomes among localized prostate cancer survivors: health-related quality-of-life changes after radical prostatectomy, external radiation, and brachytherapy. J Clin Oncol. 2005 Apr 20;23(12):2772-80. doi: 10.1200/JCO.2005.07.116. PMID 15837992
- [Background] Liu J, Mittendorf T, von der Schulenburg JM. A structured review and guide through studies on health-related quality of life in kidney cancer, hepatocellular carcinoma, and leukemia. Cancer Invest. 2010 Mar;28(3):312-22. doi: 10.3109/07357900903287022. PMID 19863345
- [Background] Somani BK, Gimlin D, Fayers P, N'dow J. Quality of life and body image for bladder cancer patients undergoing radical cystectomy and urinary diversion--a prospective cohort study with a systematic review of literature. Urology. 2009 Nov;74(5):1138-43. doi: 10.1016/j.urology.2009.05.087. Epub 2009 Sep 20. PMID 19773042
- [Background] Carpentier MY, Fortenberry JD. Romantic and sexual relationships, body image, and fertility in adolescent and young adult testicular cancer survivors: a review of the literature. J Adolesc Health. 2010 Aug;47(2):115-25. doi: 10.1016/j.jadohealth.2010.04.005. Epub 2010 Jun 11. PMID 20638003
- [Background] Kuczyk M, Machtens S, Bokemeyer C, Schultheiss D, Jonas U. Sexual function and fertility after treatment of testicular cancer. Curr Opin Urol. 2000 Sep;10(5):473-7. doi: 10.1097/00042307-200009000-00018. PMID 11005454
- [Background] Huddart RA, Norman A, Moynihan C, Horwich A, Parker C, Nicholls E, Dearnaley DP. Fertility, gonadal and sexual function in survivors of testicular cancer. Br J Cancer. 2005 Jul 25;93(2):200-7. doi: 10.1038/sj.bjc.6602677. PMID 15999104
- [Background] Matos E, Skrbinc B, Zakotnik B. Fertility in patients treated for testicular cancer. J Cancer Surviv. 2010 Sep;4(3):274-8. doi: 10.1007/s11764-010-0135-9. Epub 2010 Jul 3. PMID 20602187
- [Background] Cella D. Quality of life in patients with metastatic renal cell carcinoma: the importance of patient-reported outcomes. Cancer Treat Rev. 2009 Dec;35(8):733-7. doi: 10.1016/j.ctrv.2009.07.003. Epub 2009 Aug 21. PMID 19699588
- [Background] Carlson LE, Ursuliak Z, Goodey E, Angen M, Speca M. The effects of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients: 6-month follow-up. Support Care Cancer. 2001 Mar;9(2):112-23. doi: 10.1007/s005200000206. PMID 11305069
- [Background] Astin JA. Stress reduction through mindfulness meditation. Effects on psychological symptomatology, sense of control, and spiritual experiences. Psychother Psychosom. 1997;66(2):97-106. doi: 10.1159/000289116. PMID 9097338
- [Background] Kabat-Zinn J. Full Catastrophe Living: Using the Wisdom of your Mind to Face Stress, Pain and Illness. New York: Dell Publishing; 1990
- [Background] Bishop SR, Lau M, Shapiro S et al. Mindfulness: A Proposed Ooperational Definition. Clinical Psychology: Science and Practice 2004;11(3):230-241
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress, and immune parameters in breast and prostate cancer outpatients. Psychosom Med. 2003 Jul-Aug;65(4):571-81. doi: 10.1097/01.psy.0000074003.35911.41. PMID 12883107
- [Background] Carlson LE, Garland SN. Impact of mindfulness-based stress reduction (MBSR) on sleep, mood, stress and fatigue symptoms in cancer outpatients. Int J Behav Med. 2005;12(4):278-85. doi: 10.1207/s15327558ijbm1204_9. PMID 16262547
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress and levels of cortisol, dehydroepiandrosterone sulfate (DHEAS) and melatonin in breast and prostate cancer outpatients. Psychoneuroendocrinology. 2004 May;29(4):448-74. doi: 10.1016/s0306-4530(03)00054-4. PMID 14749092
- [Background] McDade TW, Williams S, Snodgrass JJ. What a drop can do: dried blood spots as a minimally invasive method for integrating biomarkers into population-based research. Demography. 2007 Nov;44(4):899-925. doi: 10.1353/dem.2007.0038. PMID 18232218
- [Background] Matousek RH, Pruessner JC, Dobkin PL. Changes in the cortisol awakening response (CAR) following participation in mindfulness-based stress reduction in women who completed treatment for breast cancer. Complement Ther Clin Pract. 2011 May;17(2):65-70. doi: 10.1016/j.ctcp.2010.10.005. Epub 2010 Nov 26. PMID 21457893
- [Background] Fuligni AJ, Telzer EH, Bower J, Cole SW, Kiang L, Irwin MR. A preliminary study of daily interpersonal stress and C-reactive protein levels among adolescents from Latin American and European backgrounds. Psychosom Med. 2009 Apr;71(3):329-33. doi: 10.1097/PSY.0b013e3181921b1f. Epub 2009 Feb 5. PMID 19196810
- [Background] Bankier B, Barajas J, Martinez-Rumayor A, Januzzi JL. Association between C-reactive protein and generalized anxiety disorder in stable coronary heart disease patients. Eur Heart J. 2008 Sep;29(18):2212-7. doi: 10.1093/eurheartj/ehn326. Epub 2008 Jul 4. PMID 18603621
- [Background] Bankier B, Barajas J, Martinez-Rumayor A, Januzzi JL. Association between anxiety and C-reactive protein levels in stable coronary heart disease patients. Psychosomatics. 2009 Jul-Aug;50(4):347-53. doi: 10.1176/appi.psy.50.4.347. PMID 19687175
- [Background] Bankier B, Barajas J, Martinez-Rumayor A, Januzzi JL. Association between major depressive disorder and C-reactive protein levels in stable coronary heart disease patients. J Psychosom Res. 2009 Mar;66(3):189-94. doi: 10.1016/j.jpsychores.2008.09.010. Epub 2008 Oct 9. PMID 19232230
- [Background] Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosom Med. 2009 Feb;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. Epub 2009 Feb 2. PMID 19188531
- [Background] O'Donovan A, Hughes BM, Slavich GM, Lynch L, Cronin MT, O'Farrelly C, Malone KM. Clinical anxiety, cortisol and interleukin-6: evidence for specificity in emotion-biology relationships. Brain Behav Immun. 2010 Oct;24(7):1074-7. doi: 10.1016/j.bbi.2010.03.003. Epub 2010 Mar 18. PMID 20227485
- [Background] Corwin EJ, Johnston N, Pugh L. Symptoms of postpartum depression associated with elevated levels of interleukin-1 beta during the first month postpartum. Biol Res Nurs. 2008 Oct;10(2):128-33. doi: 10.1177/1099800408323220. PMID 18829596
- [Background] Slavich GM, O'Donovan A, Epel ES, Kemeny ME. Black sheep get the blues: a psychobiological model of social rejection and depression. Neurosci Biobehav Rev. 2010 Sep;35(1):39-45. doi: 10.1016/j.neubiorev.2010.01.003. Epub 2010 Jan 18. PMID 20083138
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] GUTHRIE R, SUSI A. A SIMPLE PHENYLALANINE METHOD FOR DETECTING PHENYLKETONURIA IN LARGE POPULATIONS OF NEWBORN INFANTS. Pediatrics. 1963 Sep;32:338-43. No abstract available. PMID 14063511
- [Background] McDade TW, Stallings JF, Worthman CM. Culture change and stress in Western Samoan youth: Methodological issues in the cross-cultural study of stress and immune function. Am J Hum Biol. 2000 Nov 1;12(6):792-802. doi: 10.1002/1520-6300(200011/12)12:63.0.CO;2-F. PMID 11534070
- [Background] McDade TW, Leonard WR, Burhop J, Reyes-Garcia V, Vadez V, Huanca T, Godoy RA. Predictors of C-reactive protein in Tsimane' 2 to 15 year-olds in lowland Bolivia. Am J Phys Anthropol. 2005 Dec;128(4):906-13. doi: 10.1002/ajpa.20222. PMID 16118783
- [Background] Snodgrass JJ, Leonard WR, Tarskaia LA, McDade TW, Sorensen MV, Alekseev VP, Krivoshapkin VG. Anthropometric correlates of C-reactive protein among indigenous Siberians. J Physiol Anthropol. 2007 Mar;26(2):241-6. doi: 10.2114/jpa2.26.241. PMID 17435372
- [Background] McDade TW, Rutherford JN, Adair L, Kuzawa C. Adiposity and pathogen exposure predict C-reactive protein in Filipino women. J Nutr. 2008 Dec;138(12):2442-7. doi: 10.3945/jn.108.092700. PMID 19022970
- [Background] Mei JV, Alexander JR, Adam BW, Hannon WH. Use of filter paper for the collection and analysis of human whole blood specimens. J Nutr. 2001 May;131(5):1631S-6S. doi: 10.1093/jn/131.5.1631S. PMID 11340130
- [Background] McDade TW, Shell-Duncan B. Whole blood collected on filter paper provides a minimally invasive method for assessing human transferrin receptor level. J Nutr. 2002 Dec;132(12):3760-3. doi: 10.1093/jn/132.12.3760. PMID 12468620
- [Background] Victorson D, Hankin V, Polster R, McCurdy M, McGuire M, Brendler C. Reducing Symptoms of Anxiety for Men with Prostate Cancer on Active Surveillance and their Spouses: Initial Findings from a Randomized Clinical Trial. The Journal of Urology 2010;138(4):e180-e181
- [Background] Eyberg S, Edwards D, Boggs S, Foote R. Maintaining the Treatment Effects of Parent Training: The Role of Booster Sessions and Other Maintenance Strategies. Clinical Psychology: Science and Practice 1998;5:544-554
- [Background] Simkin-Silverman LR, Wing RR, Boraz MA, Meilahn EN, Kuller LH. Maintenance of cardiovascular risk factor changes among middle-aged women in a lifestyle intervention trial. Womens Health. 1998 Fall;4(3):255-71. PMID 9787651
- [Background] Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol. 2010 Feb;15(Pt 1):1-39. doi: 10.1348/135910709X466063. Epub 2009 Jul 28. PMID 19646331
- [Background] Kirsch NL, Shenton M, Rowan J. A generic, 'in-house', alphanumeric paging system for prospective activity impairments after traumatic brain injury. Brain Inj. 2004 Jul;18(7):725-34. doi: 10.1080/02699050310001646161. PMID 15204332
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Trapnell PD, Campbell JD. Private self-consciousness and the five-factor model of personality: distinguishing rumination from reflection. J Pers Soc Psychol. 1999 Feb;76(2):284-304. doi: 10.1037//0022-3514.76.2.284. PMID 10074710
- [Background] Roth AJ, Rosenfeld B, Kornblith AB, Gibson C, Scher HI, Curley-Smart T, Holland JC, Breitbart W. The memorial anxiety scale for prostate cancer: validation of a new scale to measure anxiety in men with with prostate cancer. Cancer. 2003 Jun 1;97(11):2910-8. doi: 10.1002/cncr.11386. PMID 12767107
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007 Dec;21(4):572-83. doi: 10.1037/0893-3200.21.4.572. PMID 18179329
- [Background] Rose M, Bjorner JB, Becker J, Fries JF, Ware JE. Evaluation of a preliminary physical function item bank supported the expected advantages of the Patient-Reported Outcomes Measurement Information System (PROMIS). J Clin Epidemiol. 2008 Jan;61(1):17-33. doi: 10.1016/j.jclinepi.2006.06.025. PMID 18083459
- [Background] Gershon R. Comparing short forms and CAT across PROMIS. 2009
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Background] Buysse DJ, Yu L, Moul DE, Germain A, Stover A, Dodds NE, Johnston KL, Shablesky-Cade MA, Pilkonis PA. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. Sleep. 2010 Jun;33(6):781-92. doi: 10.1093/sleep/33.6.781. PMID 20550019
- [Background] Clements AD, Parker CR. The relationship between salivary cortisol concentrations in frozen versus mailed samples. Psychoneuroendocrinology. 1998 Aug;23(6):613-6. doi: 10.1016/s0306-4530(98)00031-6. PMID 9802131
- [Background] Kirschbaum C, Wolf OT, May M, Wippich W, Hellhammer DH. Stress- and treatment-induced elevations of cortisol levels associated with impaired declarative memory in healthy adults. Life Sci. 1996;58(17):1475-83. doi: 10.1016/0024-3205(96)00118-x. PMID 8622574